CLINICAL TRIAL: NCT02769546
Title: Physician-Patient Communication and Expectations Regarding Ovarian Cancer Prognosis
Status: Terminated | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 28815
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Surveys

SUMMARY:
The primary objective is to administer a cross-sectional survey to directly compare the differences patients and physicians hold regarding ovarian cancer prognosis and survival, complications arising from treatment, and counseling on advance directives, living wills, palliative care, and hospice services. Overall, the project will pinpoint opportunities for better patient physician communication regarding prognosis and end-of-life care and allow for more informed and tailored decision-making.

ELIGIBILITY:
Inclusion Criteria:

* women over 18 years old with biopsy-confirmed malignancy
* being actively treated or are in surveillance for epithelial ovarian cancer
* have an existing therapeutic relationship with a provider who is participating in the study.

Exclusion Criteria:

* patients enrolled in palliative or hospice care programs, patients with a second primary malignancy within the last five years (excluding non-melanoma skin cancer)
* patients who are illiterate or non-English speaking, and patients without decision-making capacity.
* There are no exclusion criteria based on age, gender, economic status or race/ethnicity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian Cancer
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of completed surveys and phone interviews | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Haggerty, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States